CLINICAL TRIAL: NCT03705975
Title: Randomized Controlled Trial, Manual Treatment and Classical Physiotherapy for One Group, PNF and Classical Physiotherapy for Other Group
Brief Title: Manual Treatment and Proprioceptive Neuromusculer Fasilitation Techniques for Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Canli, research assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Filiz Can
Record Dates: First submitted 2018-09-19; First posted 2018-10-15 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-06

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edit arms (Active Comparator): classical physiotherapy and manual treatment. Classical physiotherapy consisting of hotpack and ultrason. Hotpack duration is 20 minutes and ultrason duration is 5 minutes in one session. Manual treatment is consist of scapular mobilization, glenohumeral joint inferior and posterior mobilization. Treatment modality is implemented by physical therapist three times a week for 8 weeks.
  Interventions: Other: Manual treatment
- edit arm/intervention cross (Active Comparator): classical physiotherapy and proprioceptive neuromusculer fasilitation. Classical physiotherapy consist of hotpack and ultrason. Hotpack duration is 20 minutes and ultrason duration is 5 minutes in one session. Scapular PNF and upper extremity PNF (flexion-abduction-external rotation) pattern. Treatment programme was implemented by physical therapist three times a week for 8 weeks.
  Interventions: Other: Manual treatment

INTERVENTIONS:
Other: Manual treatment — Scapula mobilization, glenohumeral joint mobilization

SUMMARY:
This study aim was to compare the effectiveness of manual treatment and proprioceptive neuromuscular fasilitation (PNF) techniques in patients with adhesive capsulitis. One group will receive classical physical therapy including hotpack,ultrason and in additon manual treatment application. Other group receive classical physical therapy including hotpack, ultrason and in addition PNF techniques. Two group will be made wand exercise at home three times a day 10 times at one session.

DETAILED DESCRIPTION:
There is no consensus physical therapy treatment protocol in adhesive capsulitis. It is because it etiology and pathophysiology is unknown. Also it has different clinical stage. PNF techniques often used by physical therapist in adhesive capsulitis aim increasing range of motion, improving muscle strenght and decreasing pain. PNF techniques improves neuromusculer control of central nervous system via stimulating muscle spindles, golgi tendon organs and other receptors in connective tissue. However, there is limited evidence effectivenes of PNF techniques in adhesive capsulitis.

Other technique often used by physical therapist in adhesive capsulitis is manual treatment. Manual treatment decreases pain and improves function. It re-arrange glenohumeral joint arthrocinematic. It diminishes capsule fibrosis.

There is no reasearh aimed comparing the PNF and manual treatment. Our aim was to compare the effectiveness of manual treatment and PNF techiques in patients with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* adhesive capsulitis due to idiopathic or acquired reasons

Exclusion Criteria:

* Cervical disk hernia
* Neuromusculer disease
* Shoulder impingement syndrome
* Rotator cuff tear
* Corticosteroid enjeksion in shoulder
* Tumour
* Physical therapy or manual treatment is implemented same shoulder last 6 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-18 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Range of motion change | change from baseline range of motion assessment at 8 weeks
  Flexion, abduction, internal and external rotation range of motion will assessed with universal goniometer.

SECONDARY OUTCOMES:
Subjective pain assessment: VAS | Change from baseline subjective pain assessment at 8 weeks
  Rest, activity and night pain will be assessed by Visuel Analog Scale (VAS). It is self reported pain scale.We will question the intensty of shoulder region pain at rest, night and activity by VAS. The pain intensity was scored on a 100-mm visual analog scale (VAS) where 0 cm indicated "no pain" and 10 cm indicated "worst imaginable pain.
Scapular dyskinesis | Change from baseline scapular dyskinesis assessment at 8 weeks
  Scapular dyskinesis will be assessed with Lateral Scapular Slide Test. To measure we used tape measure.
Muscle strenght | Change from baseline muscle strenght assessment at 8 weeks
  Shoulder complex muscle strenght will be assssed by muscle dynamometer.
General arm function | Change from baseline shoulder function assessment at 8 weeks
  Shoulder function will be assessed using Disabilities of the Arm, Shoulder and Hand Questionnare (DASH),
Health quality depent on health | Change from baseline health quality assessment at 8 weeks
  Health quality depent on health will be assessed using the "Quality of Life (SF-36)" questionnare. Assesses 8 dimensions of health with 36 items such as physical function, social function, role constraints, mental health, vitality (energy), pain and general perception of health. Each subsection of the quality of life questionnaire is scored between 0 and 100 points. Higher score indicates better outcome.
Health quality is not related to health | Change from baseline health quality assessment at 8 weeks
  Health quality is not related to health will be assessed using the " World Health Organization Quality of Life Assessment (EUROHIS-QOL)". It contains 8 questions. Two of the questions include general health and general quality of life questions, while the remaining 6 questions consist of questions about physical, spiritual, environmental and social dimensions.These questions how long the patient has experienced some things in the last two weeks, what they can do, whether it is good or satisfying, what they think about the quality of life, health and other aspects of life. The total score is calculated by summing the items. The total score is between 8 and 40 points. Higher score indicate worse outcome.
general health level | Change from baseline general health level assessment at 8 weeks
  general healt level will be assessed using "Health Assessment Questionnaire". Health Assessment Questionnare two to three questions in each of eight areas of activities of daily living (ADL): dressing and grooming, arising. eating, walking, hygiene, reach, grip, and activities. The total score ranges between 0-24. The highest score indicate more disability level.
Self rated upper extremity disablity and symptoms. | Change from baseline general health level assessment at 8 weeks
  Self rated upper extremity disablity and symptoms will be assessed using the "Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH)" survey. 30 items (total score): 6 items about symptoms (3 about pain, 1 for tingling/numb-ness, 1 for weakness, 1 for stiffness) and 24 about function (21 about physical function, 3 about social/role function). The patients point out the appropriate response between 1-5 points according to the Likert system for each question (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: no disability). A score of 0-100 points is obtained from each section according to the results of the DASH survey ( 0=no disability, 100=most severe disability). 0 score indicate best and 100 score indicate worst outcome. Higher values represent worse outcome.
Self-assessment of symptoms and function of the shoulder | Change from baseline general health level assessment at 8 weeks
  Self-assessment of symptoms and function of the shoulder will be assessed using the Shoulder Pain and Disability Index (SPADI).The SPADI total score is the unweightedmean of the pain and function subscores.Originally, 0 score indicate best and 100 score indicate worst.
To assess functional disability of the shoulder | Change from baseline general health level assessment at 8 weeks
  Functional disability of the shoulder will be assessed using the Simple Shoulder Test.Total score of 12 items: 2 about function related to pain, 7 about function/strength,and 3 about range of motion.0 score indicate worst and 100 score indicate best function.

CONTACTS AND LOCATIONS:
Locations (1):
- Kübra, Ankara, Sıhhıye, Turkey (Türkiye)